CLINICAL TRIAL: NCT02797951
Title: A Phase 3b Multicenter, Single-Arm, Open-Label Safety Study of LY2951742 (Galcanezumab) in Patients With Episodic or Chronic Cluster Headache
Brief Title: A Study of LY2951742 (Galcanezumab) in Participants With Cluster Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16351; I5Q-MC-CGAR (Other: Eli Lilly and Company); 2015-005234-21 (EudraCT Number)
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Results first posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Episodic Cluster Headache; Chronic Cluster Headache
Keywords: cluster headache; headache; brain diseases; central nervous system diseases; headache disorders; headache disorders, primary; nervous system diseases; neurologic manifestations; pain; trigeminal autonomic cephalalgias
MeSH Terms: conditions — Cluster Headache; Headache; Brain Diseases; Central Nervous System Diseases; Headache Disorders; Headache Disorders, Primary; Nervous System Diseases; Neurologic Manifestations; Pain; Trigeminal Autonomic Cephalalgias | interventions — galcanezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Galcanezumab (Experimental): Participants received 300 milligram (mg) Galcanezumab administered subcutaneously (SC) up to once a month.
  Interventions: Drug: Galcanezumab

INTERVENTIONS:
Drug: Galcanezumab — Administered SC
  Other Names: LY2951742

SUMMARY:
The main purpose of this study is to assess the long-term safety and tolerability of galcanezumab administered up to once monthly in participants with episodic or chronic cluster headache who have completed study I5Q-MC-CGAL (NCT02397473) or study I5Q-MC-CGAM (NCT02438826).

ELIGIBILITY:
Inclusion Criteria:

* Participants who participated in and completed either study CGAL or study CGAM.
* Investigator judges the participant as reliable to follow all study procedures, keep all study visits, and be compliant with study requirements.

Exclusion Criteria:

* Current enrollment in or discontinuation within the last 30 days from, a clinical trial involving any investigational drug or device (with the exception of Study CGAL or Study CGAM).
* Current use or any prior exposure to any calcitonin-gene-related peptide (CGRP) antibody, any antibody to the CGRP receptor, or antibody to nerve growth factor (NGF) (with the exception of Study CGAL or Study CGAM).
* A history of migraine variants that could implicate or could be confused with ischemia.
* Known hypersensitivity to multiple drugs, monoclonal antibodies or other therapeutic proteins.
* A history or presence of other medical illness that indicates a medical problem that would preclude study participation.
* Evidence of significant active or unstable psychiatric disease, in the opinion of the investigator.
* Women who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (40):
- United States (11):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Stanford University Hospital, Palo Alto, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Colorado Neurological Institute, Englewood, Colorado
  - New England Institute for Clinical Research, Stamford, Connecticut
  - University of South Florida, Tampa, Florida
  - Atlanta Center of Medical Research, Atlanta, Georgia
  - Michigan Head, Pain and Neurological Institute, Ann Arbor, Michigan
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Northwest Clinical Research Center, Bellevue, Washington
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - Centre Hospitalier Regional de la Citadelle, Liège
- Canada (2):
  - Stroyan Research, Toronto, Ontario
  - Centre de Traitement Neurologique, Montreal
- Glostrup Hospital, Glostrup Municipality, Denmark
- Finland (2):
  - Suomen Terveystalo, Jyväskylä
  - Terveystalo Pulssi, Turku
- France (5):
  - CHRU de Lille - Hôpital Roger Salengro, Lille, Cedex
  - APHM Hôpital de la Timone, Marseille
  - Hôpital de Cimiez, Nice
  - Hopital Lariboisière, Paris
  - CHU St Etienne Hopital Nord, Saint-Etienne
- Germany (5):
  - Klinikum der Universität München, München, Bavaria
  - Migräne- und Kopfschmerzklinik GmbH & Co. KG, Königstein im Taunus, Hesse
  - Praxis Dr. Philipp Stude, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Jena, Jena, Thuringia
  - Universitaetsklinikum Essen, Essen
- Greece (2):
  - 401 Army General Hospital of Athens, Athens, Attica
  - Eginition Hospital of Athens, Athens
- Italy (3):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Istituto Neurologico Carlo Besta, Milan
  - Fondazione Istituto Neurologico Nationale C. Mondino, Pavia
- Netherlands (2):
  - Boerhaave Medisch Centrum, Amsterdam
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínico Universitario de Valencia, Valencia
- United Kingdom (3):
  - Hull Royal Infirmary, Hull, East Yorkshire
  - Walton Centre for Neurology and Neurosurgery, Liverpool, Lancashire
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Riesenberg R, Gaul C, Stroud CE, Dong Y, Bangs ME, Wenzel R, Martinez JM, Oakes TM. Long-term open-label safety study of galcanezumab in patients with episodic or chronic cluster headache. Cephalalgia. 2022 Oct;42(11-12):1225-1235. doi: 10.1177/03331024221103509. Epub 2022 May 27. PMID 35633025
- See also: A Study of LY2951742 (Galcanezumab) in Participants With Cluster Headache — https://trials.lillytrialguide.com/en-US/trial/WEzAu0Rzqgg2YY8AKeKSC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed one of the parent studies I5Q-MC-CGAL (NCT02397473) or I5Q-MC-CGAM (NCT02438826) were enrolled in this study.
Groups:
- Galcanezumab 300 mg SC: Participants received 300 milligram (mg) Galcanezumab administered subcutaneously (SC) up to once a month.
Period: Overall Study
Arm/Group | Galcanezumab 300 mg SC
Started | 165
Received at Least One Dose of Study Drug | 164
Completed (Participants who continued until sponsor ended the study following regulatory approval or non-approval of study drug for cluster headache indication in a country/region.) | 116
Not Completed | 49
Not completed — Adverse Event | 4
Not completed — Death | 1
Not completed — Lack of Efficacy | 19
Not completed — Lost to Follow-up | 4
Not completed — Physician Decision | 6
Not completed — Withdrawal by Subject | 15

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Galcanezumab 300 mg SC: Participants received 300 mg Galcanezumab administered SC up to once a month.
Arm/Group | Galcanezumab 300 mg SC
Number analyzed (Participants) | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.30 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 117
  Unknown or Not Reported | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 140
  More than one race | 19
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 17
  Canada | 7
  Denmark | 4
  Finland | 5
  France | 23
  Germany | 25
  Greece | 2
  Italy | 24
  Netherlands | 8
  Spain | 17
  United Kingdom | 4
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious AEs (SAEs)
Description: A TEAE is defined as the reported AEs that first occurred or worsened during the post-baseline phase compared with the baseline phase.
  An SAE is any adverse event from this study that results in 1 of the following: Death, initial or prolonged inpatient hospitalization, a life-threatening experience (that is, immediate risk of dying), persistent or significant disability/incapacity, congenital anomaly/birth defect, Important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent 1 of the other outcomes listed in the definition above. A summary of serious and other non-serious adverse events regardless of causality is located in the reported adverse events module.
Time Frame: Baseline through End of Study (Up to 4 Years)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Galcanezumab 300 mg SC
Number analyzed (Participants) | 164
Participants
  TEAEs | 119
  SAEs | 17

2. Primary Outcome: Number of Participants With Suicidal Ideation and Behaviours Collected by Columbia - Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a scale capturing occurrence, severity, and frequency of suicide-related thoughts and behaviours, and has a binary response (yes/no).
  * Suicidal Ideation: a "yes" answer to any one of 5 suicidal ideation questions: Wish to be Dead, Non-specific Active Suicidal Thoughts, Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act, Active Suicidal Ideation with Some Intent to Act, without Specific Plan, Active Suicidal Ideation with Specific Plan and Intent.
  * Suicidal Behaviour: a "yes" answer to any of 5 suicidal behaviour questions: Preparatory Acts or Behaviour, Aborted Attempt, Interrupted Attempt, Actual Attempt (non-fatal), Completed Suicide.
Time Frame: Baseline through End of Study (Up to 4 Years)
Population: All participants who received at least one dose of study drug and had at least one postbaseline C-SSRS assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Galcanezumab 300 mg SC
Number analyzed (Participants) | 164
Participants
  Suicidal Ideation | 2
  Suicidal Behaviour | 0

3. Secondary Outcome: Number of Participants With Treatment Emergent Anti-Drug Antibodies (TE-ADA) to Galcanezumab
Description: A participant is considered TE-ADA positive if:
  * ADA "not present" baseline result and any subsequent "present" postbaseline ADA result with a titer of at least 1:20 (treatment-induced), or
  * ADA "present" baseline result and any subsequent "present" postbaseline ADA result with a 4-fold or greater increase in titer from baseline (treatment-boosted).
Time Frame: Baseline through End of Study (Up to 4 Years)
Population: All participants who received at least one dose of study drug and had baseline and at least one post baseline ADA assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Galcanezumab 300 mg SC
Number analyzed (Participants) | 159
Participants | 8

ADVERSE EVENTS:
Time Frame: Baseline through End of Study (Up to 4 Years)
Description: All participants who received at least one dose of study drug.
Arm/Group | Galcanezumab 300 mg SC
All-Cause Mortality (participants affected / at risk) | 1/164
Serious Adverse Events (participants affected / at risk) | 17/164
Other Adverse Events (participants affected / at risk) | 62/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galcanezumab 300 mg SC (N=164)
Constipation (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1)
Exposure to household chemicals (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cluster headache (Nervous system disorders) | 3 (3)
Sciatica (Nervous system disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) — This event was not captured in the C-SSRS suicidal behaviour count as the participant's responses to suicidal ideation/behaviours were "no" for all completed assessments.
Ureterolithiasis (Renal and urinary disorders) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galcanezumab 300 mg SC (N=164)
Bronchitis (Infections and infestations) | 10 (16)
Influenza (Infections and infestations) | 16 (21)
Nasopharyngitis (Infections and infestations) | 36 (46)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT02797951/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT02797951/SAP_001.pdf